CLINICAL TRIAL: NCT07113444
Title: The Acute Effect of Tai Chi Versus Moderate-Intensity Combined Exercise on Cardiovascular, Metabolic, and Cardiac Autonomic Control Parameters in Older Men and Women With Type 2 Diabetes Mellitus: A Randomized, Single-Blind, Crossover Controlled Trial
Brief Title: Acute Effect of Tai Chi Versus Moderate-Intensity Combined Exercise on Cardiovascular, Metabolic, and Cardiac Autonomic Control Parameters in Older Men and Women With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Emmanuel Gomes Ciolac, Full Professor of Department of Physical Education, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 88582225.1.0000.5398
Record Dates: First submitted 2025-07-22; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: Tai Ji; Diabetes Mellitus, Type 2; Blood Glucose; Cross-Over Studies; Vascular Stiffness; Endothelium, Vascular
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Crossover Model (All participants will get all interventions in random order: Tai Chi, MICE, and control.)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): 40-60 minute supervised Yang-style Tai Chi lesson (24-form simplified pattern). Focus on calm, controlled movements and breathing coordination.
  Interventions: Other: Tai Chi
- Moderate-Intensity Exercise (MICE) (Experimental): The MICE session will consist of five minutes of warm-up (joint mobility and stretching exercises between PSE levels 9 and 11, 30 minutes of walking on the treadmill between PSE levels 12 and 13, 20 minutes of muscle strengthening exercises between levels 12 and 14 of PSE (two sets of 15 to 20 repetitions in circuit in the exercises bent row with elastic band, bodyweight squats, adapted push-ups (on the wall or on the counter), deadlifts with an elastic band, presses with an elastic band and an abdominal band on the floor or adapted on the chair) and five minutes of back to calm (light stretching and breathing exercises at PSE level 9).
  Interventions: Other: Moderate-Intensity Combined Exercise (MICE)
- Control (No Exercise) (Sham Comparator): The CON session will consist of 60 minutes of rest in the sitting position. Participants will be told not to sleep and will not have access to reading or electronic devices during the CON session.
  Interventions: Other: Control ( No Exercise )

INTERVENTIONS:
Other: Tai Chi — Yang style of Tai Chi (24 form)
  Other Names: Tai ji; Tai Chi Chuan
  Arms: Tai Chi
Other: Moderate-Intensity Combined Exercise (MICE) — start from warm up (5 minute )repetitions in circuit in the exercises bent row with elastic band, bodyweight squats, adapted push-ups (on the wall or on the counter), deadlifts with an elastic band, presses with an elastic band and an abdominal band on the floor or adapted on the chair and cool down in the end
  Arms: Moderate-Intensity Exercise (MICE)
Other: Control ( No Exercise ) — The CON session will last 60 minutes and will be conducted only sitting. Participants will be told not to sleep and will not be allowed to use reading materials or any electrical gadgets during the CON session.
  Arms: Control (No Exercise)

SUMMARY:
Type 2 diabetes mellitus (T2DM) in the elderly population is associated with compromised cardiovascular and metabolic functions, thereby necessitating the implementation of safe exercise interventions. This study employs a randomized, single-blind, crossover design will be conducted in Brazil to examine whether Tai Chi, a low-impact mind-body exercise, offers acute benefits comparable to those of moderate-intensity combined exercise (MICE) in 24 older adults (≥65 years) diagnosed with T2DM, consisting of 12 men and 12 women. Participants recruited through community advertisements and screened to ensure inactivity, stable medication usage, and the absence of significant comorbidities will undergo randomized sessions of Tai Chi, MICE, and a control (CON) intervention. Evaluations will include capillary blood glucose (the primary outcome), blood pressure, heart rate variability, arterial stiffness (PWVcf), and endothelial function (FMD) measured before, immediately after, and 45minute post-intervention, along with 24-hour ambulatory monitoring. Standardized protocols will be employed to regulate physical activity. By juxtaposing these interventions, the study seeks to ascertain if Tai Chi could serve as a feasible alternative for enhancing acute metabolic and cardiovascular responses in older diabetic adults, thus providing practical insights for clinical and lifestyle management.

ELIGIBILITY:
Inclusion Criteria:

only with type 2 diabetes

Exclusion Criteria:

* if not able to perform physical exercise (Extreme neuropathy, wounds in the feet, and amputation risk.)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Capillary blood glucose change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Capillary blood glucose will be measured using a digital glucometer (FreeStyle Optium Neo, 163 Abbott, Oxon, UK) in milligrams per deciliter (mg/dL)

SECONDARY OUTCOMES:
Carotid-femoral pulse wave velocity (PWVcf) change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Carotid-femoral pulse wave velocity (PWVcf) will be measured using an automated device (Complior Analyze™ PWV and Central Pressure Analysis™; AlamMedical, Saint-Quentin-Fallavier, France), in meters per second (m/s)
Brachial artery flow-mediated dilation (FMD) change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Brachial artery flow-mediated dilation (FMD) will be measured using an ultrasound device (SonoSite M-Turbo™; Fujifilm Inc., Bothell, Washington, USA), and will consist in the brachial artery diameter difference between before (baseline diameter) and after (peak diameter) the artery occlusion for 5 minutes. FMD will be expressed in percentage (%) and will be determined by the following formula: FMD (%) = (peak diameter - baseline diameter)/baseline diameter × 100
Central blood pressures change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Central blood pressures will be assessed directly from the carotid pressure waveform, in millimeters of mercury (mmHg), and using a non-invasive automated device (Complior Analyze™ PWV and Central Pressure Analysis™; AlamMedical, Saint-Quentin-Fallavier, France)
Heart rate variability (HRV) change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Heart rate variability will be assesseded using a digital telemetry system (Polar H10™, Polar Electro Inc, Kempele, Finland) to measure HR signals beat-to-beat. A sequence of 256 stable R-R intervals will be used to calculate frequency and time domain indexes, in hertz (Hz) and milliseconds (ms), respectively
Brachial blood pressure (BP) change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Systolic and diastolic brachial blood pressure (BP) will be measured using an automatic monitor (Omron HEM 7200™, Omron Healthcare Inc., Dalian, China) in millimeters of mercury (mmHg)
24-hour ambulatory blood pressure monitoring (ABPM) difference between interventions | 24 hours
  Ambulatory systolic and diastolic blood pressure monitoring (ABPM), in millimeters of mercury (mmHg), will be measured for 24 hours after the end of each visit (approximately 90 minutes after the end of the Tai Chi, moderate-intensity combined exercise and control interventions), after a brief bath and using an automatic equipment (CardioMapa™, Cardios Sistemas Comercial e Industrial Ltda., São Paulo, Brazil).
24-hour heart rate variability (HRV) difference between interventions | 24 hours
  Ambulatory heart rate variability (HRV) will be assessed for 24 hours after the end of each visit (approximately 90 minutes after the end of the Tai Chi, moderate-intensity combined exercise and control interventions), after a brief bath and using an automatic equipment (CardioMapa™, Cardios Sistemas Comercial e Industrial Ltda., São Paulo, Brazil). The will measure the heart rhythm (3-lead electrocardiogram), and the R-R intervals will be used to calculate frequency and time domain indexes, in hertz (Hz) and milliseconds (ms), respectively

OTHER OUTCOMES:
Augmentation Index (AIx) change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Derived from central pressure waveforms via Complior Analyze™. Calculated as: [(Second systolic peak - First systolic peak) / Pulse pressure] × 100. Reported in %.
Heart rate change from baseline | Baseline (minute 0), immediately after the intervention (minute 60) and 45 minutes after the intervention (minute 105)
  Heart rate will be measured using a digital telemetry system (Polar H10™, Polar Electro Inc, Kempele, Finland) in beats per minute (bpm)

IPD SHARING:
Plan to Share IPD: Yes
Participants who are interested in participating will provide an anamnesis to the investigator. The investigator will evaluate the IDP eligibility or non-eligibility criteria. Each qualified participant will get a document that includes the research protocol, statistical analysis plan, informed consent form, clinical study report, and analytic code information. Thus, scientists will do cardiopulmonary activity tests to assess if IDP will be able to study the program.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Initial data will be analysed after completing all 3 interventions .
Access Criteria: Informed Consent Form described and signed. DP will received Informed Consent Form informing the objectives, study deling, interventions, analyses, risks and benefits. Participation in this study will be voluntary and confidential after signing of an informed consent.
URL: https://plataformabrasil.saude.gov.br/